CLINICAL TRIAL: NCT02247895
Title: Effect of Treatment With the Niveus Medical Muscle Stimulation System 110 on Quadriceps Strength In Mechanically Ventilated Patients
Brief Title: Treatment of Muscle Weakness in Critically Ill Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty meeting enrollment goals
Sponsor: Gerald Supinski (Other)
Responsible Party: Sponsor-Investigator, Gerald Supinski, Staff Physician, Division of Pulmonary, Critical Care and Sleep Medicine, Principal Investigator, Professor of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 062014; 14-0237-F3R (Other: University of Kentucky)
Record Dates: First submitted 2014-09-02; First posted 2014-09-25 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Critical Illness; Respiratory Failure; Myopathy; Weakness
Keywords: ICU Acquired weakness; Critical illness; Mechanical ventilation
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency; Muscular Diseases; Asthenia | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham Treatment (Sham Comparator): Sham stimulation twice daily
  Interventions: Device: Sham Treatment
- Active Treatment (Active Comparator): The active treatment group will receive neuromuscular electrical stimulation to both quadriceps muscle for 30 minutes twice daily for a total of 14 treatments.
  Interventions: Device: Electrical stimulation

INTERVENTIONS:
Device: Sham Treatment — Subjects will undergo the same protocol as the treatment group except no electrical stimulation will be applied.
  Other Names: Sham treatment without electrical stimulation
  Arms: Sham Treatment
Device: Electrical stimulation — Two thirty minute sessions of neuromuscular electrical stimulation applied to both quadriceps for seven days for a total of 14 treatments
  Arms: Active Treatment

SUMMARY:
Patients who are admitted to the intensive care unit and require mechanical ventilation frequently develop profound respiratory and limb muscle weakness. Studies show that the development of weakness during the ICU stay results in poor outcomes. Currently there are no treatments for this muscle weakness, but it has been suggested that this weakness might improve with physical therapy. Electrical stimulation is a method to provide direct stimulation to the muscles potentially enhancing function and improving strength. The purpose of this study is to test the hypothesis that neuromuscular electrical stimulation of the quadriceps muscle will improve muscle strength in patients who are critically ill on mechanical ventilation.

DETAILED DESCRIPTION:
The basic study design is to:

1. Obtain informed consent from patient or the patients LAR
2. Randomize subjects to treatment with either:

   1. Sham therapy, consisting of bilateral placement of Niveus Medical Muscle Stimulation System 110 electrodes for 30 minutes twice daily without activation of the electrical circuitry of the unit, or
   2. Active therapy, using the Niveus Medical Muscle Stimulation System 110 electrodes to actively produce a rhythmic quadriceps contraction for 30 minutes twice daily
3. Measure magnetic stimulated quadriceps twitch (QuadTw) strength bilaterally as well as ultrasound assessment of quadriceps size
4. Continue sham or active treatment daily for 7 days for a total of 14 sessions
5. Repeat measurements of magnetic stimulated QuadTw strength and ultrasound assessment of quadriceps size on Day 8 or before Day 8 if the subject is to be discharged from the hospital prior to the allotted duration of sham or active treatment
6. Functional measurement of the patient using the Functional Status Score for the ICU (FSS-ICU) at the end of the treatment period or upon discharge
7. A member of the research team will visit the subject until hospital discharge and will record total duration (days) of mechanical ventilation, duration (days) of mechanical ventilation following study entry, duration of ICU stay, ventilator weaning time (days measured from time of first spontaneous breathing trial to extubation), and total duration (days) of hospitalization
8. The investigators will also review each subject's medical record on entry into the study to obtain demographic information including the following: age, sex, diagnoses, medications, reason for institution of mechanical ventilation, vital signs at the time of the initial visit, bedside parameters of mechanical ventilation use (including mode of ventilation, duration of ventilation, level of oxygen, breath volume and rate, % triggered breaths), most recent arterial blood gas values, and chest radiograph readings at the time of the initial visit. The investigators will also record the subject's weight, BMI and total intake and output values since admission to the ICU. In addition, investigators will monitor each subject's progress in the ICU daily by reviewing the subject's medical record and recording the clinical parameters as well as recording daily weights and total intake and output. These parameters will also be assessed until the time that the patient is discharged from the ICU. In addition, the investigators will record and note all physical therapy and occupational therapy sessions that the subject receives as part of the standard of care in the ICU and in the hospital up until the time of discharge. In the University of Kentucky hospital, occupational therapy records the Barthel Index at each session which uses a scale of 0-100 to assess an individual's functional independence when performing activities of daily living (ADLs). Physical therapy assesses functional status using Kansas University Hospital Physical Therapy Acute Care Functional Outcomes, which also assesses functional status in the categories of bed mobility, transfer, gait and walking distance.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure requiring mechanical ventilation

Exclusion Criteria:

* Attending physician on service determines that patient too unstable to tolerate measurements
* Patient requires > 15mcg/min norepinephrine or > 15mg/kg/min of dopamine.
* Fraction of inspired oxygen > 80% or positive end expiratory pressure > 15 cm H20 requirements.
* Cardiac pacemaker or implanted defibrillator.
* Neuromuscular blocking agents delivered within 48 hours of preceding testing.
* Existing neuromuscular disease.
* Profound uncorrectable hypokalemia (< 2.5) OR hypophosphatemia (< 1.0)
* Acute lower extremity deep vein thrombosis
* Pregnancy
* Prisoner
* Institutionalized patient
* If primary attending determines that patient is terminal and will likely have care withdrawn within 7 days
* Do not resuscitate order
* Body mass index > 40
* Patients requiring mechanical ventilation more than 4 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Technical Feasibility, that is ability to complete therapy sessions | Discharge from ICU, Average 7-10 days
  Percentage of patients who completed treatment with the device

SECONDARY OUTCOMES:
Total ICU length of stay | Discharge from ICU, Average 7-10 days
  Average 7-10 days
Hospital Length of Stay | Hospital discharge, Average 14-21 days
  Average 14-21 days
Functional Status Score for ICU | ICU discharge, Average 7-10 days after study entry
  Average 7-10 days after study entry
Duration of mechanical ventilation after study entry | Until patient is successfully weaned from mechanical ventilation, Average 4-10 days
  Average 4-10 days
Change in quadriceps twitch force generation | Baseline (prior to Treatment) and Day 8
  Quadriceps twitch force generation will be measured using magnetic stimulation of each femoral nerve and compared to measurements obtained at the time of study entry (baseline-prior to randomization)

OTHER OUTCOMES:
Rectus Femorus thickness | Day 8
  Rectus femorus thickness will be measured using ultrasound at baseline (study entry) and on Day 8 of study after either sham treatment or neuromuscular stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S. Supinski, MD, Principal Investigator — Professor of Medicine
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States